CLINICAL TRIAL: NCT01219062
Title: Comparative of Postoperative Pain Control at 24 and 48 Hours Between Intrathecal 0.1 mg. of Morphine or Local Infiltration of 20 ml. of 0.25% Bupivacaine in Patients Post Hip Hemiarthroplasty Under Spinal Anesthesis
Brief Title: Postoperative Pain Control After Hip Hemiarthroplasty: Intrathecal Morphine vs Periarticular Infiltration of Bupivacaine
Status: Terminated | Phase: Phase 4 | Type: Interventional
Why Stopped: Surgeon team were not happy with the study protocol, the periarticular injection of local anesthetics
Sponsor: Mahidol University (Other)
Responsible Party: Principal Investigator, Aphichat Suphathamwit,, Lecturer, Mahidol University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: Si391/2010
Record Dates: First submitted 2010-09-15; First posted 2010-10-13 (Estimated); Last update posted 2016-10-04 (Estimated); Status verified 2016-10

CONDITIONS: Femoral Neck Fracture
MeSH Terms: conditions — Femoral Neck Fractures | interventions — Morphine; Bupivacaine

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (3):
- control (Placebo Comparator): The patient will be performed spinal anesthesia alone, with postoperative PCA
  Interventions: Other: control
- Morphine (Active Comparator): The patient will received intrathecal Morphine for 0.1 mg. in Isobaric bupivacaine in spinal anesthesia and postoperative PCA
  Interventions: Drug: morphine
- bupivacaine (Active Comparator): the patients will be received spinal anesthesia and periarticular tissue infiltration with 0.25% Bupivacaine and postoperative pain control by IV PCA
  Interventions: Drug: Bupivacaine

INTERVENTIONS:
Drug: morphine — periarticular infiltration with 0.25% Bupivacaine for 20 ml.
  Arms: Morphine
Other: control — the patients will be received spinal anesthesia with 0.5% Isobaric Bupivacaine and postoperative pain control by intravenous (IV) Patient - control Analgesia (PCA)
  Arms: control
Drug: Bupivacaine — the patients will be received spinal anesthesia and periarticular tissue infiltration with 0.25% Bupivacaine and postoperative pain control by IV PCA
  Arms: bupivacaine

SUMMARY:
Falls are a common problem in elderly people which they have to receive the operation. Hemiarthroplasty is one of the common orthopedics operations. The prompt operation and good pain control will provide the good recovery and outcome. The investigators compare the efficacy of postoperative pain control between Intrathecal morphine 0.1 milligrams (mg.) with the local infiltration of 0.25% Bupivacaine for 20 milliliters (ml.) in patients received hip hemiarthroplasty under spinal anesthesia.

DETAILED DESCRIPTION:
Study process All the patients who assigned the hip hemiarthroplasty without any exclusion criteria will be enrolled in the study and be divided into 3 groups randomly

1. control group : the patients will be received spinal anesthesia with 0.5% Isobaric Bupivacaine and postoperative pain control by intravenous (IV) Patient - control Analgesia (PCA)
2. Morphine group : the patients will be received 0.1 mg. of Morphine added in Isobaric Bupivacaine for spinal anesthesia and postoperative pain control by IV PCA
3. Local group : the patients will be received spinal anesthesia and periarticular tissue infiltration with 0.25% Bupivacaine and postoperative pain control by IV PCA

Data collection

1. Demographic data : age, sex, Body Weight, Body Mass Index (BMI), ...
2. Pain score every 3 hours postoperatively in the first 6 hours and at the 12th hours by visual analogue scoring system
3. Patient global assessment and patient satisfactory visual analogue scoring system at 24th and 48th hour
4. the amount of morphine during 24 and 48 hours postoperative and the time of first dose they received

ELIGIBILITY:
Inclusion Criteria:

* age between 18-90 years
* Co-operative, able to use PCA
* ASA classification 1-3
* no contraindication for Spinal Anesthesia
* patient acceptance for spinal anesthesia
* body weight > 30 kg.
* BMI between 20-35
* no history of drug allergy, e.g. Local Anesthetics, Paracetamol, etc.

Exclusion Criteria:

* age > 90 years
* previous Hemiarthroplasty (the same site)
* pathological fracture such as severe infection, bone cancer

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2010-09; Primary Completion 2011-04 (Actual); Study Completion 2011-04 (Actual)

PRIMARY OUTCOMES:
The Amount of Morphine consumption after Hemiarthroplasty | 24 hours

SECONDARY OUTCOMES:
Efficacy of pain control | 48 hours
  Efficacy of pain control measured by
  * the amount of morphine which the patient needed to keep pain score 2-3
  * patient global assessment
  * patient satisfaction assessed by visual analogue scale
  * incidence of adverse effect such as pruritus, nausea and vomiting,...

CONTACTS AND LOCATIONS:
Overall Officials: Thitima Chinachoti, MD, Principal Investigator — Siriraj Hospital
Locations (2):
- Thailand (2):
  - Faculty of Medicine Siriraj Hospital, Bangkok
  - Thitima Chinachot, Bangkok